CLINICAL TRIAL: NCT05526703
Title: A Randomized, Double-blind, Multi-center, Therapeutic Confirmatory, Phase 3 Trial To Evaluate the Efficacy and Safety of D064 and D701 Combination Therapy in Essential Hypertension Subjects Inadequately Controlled by D064 Monotherapy
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of D064 and D701 Combination Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A30_14HT2209
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Drug: D064, D701, placebo of D012
- Comparator Group (Active Comparator)
  Interventions: Drug: D012, placebo of D064, placebo of D701

INTERVENTIONS:
Drug: D064, D701, placebo of D012 — Experimental Group Subjects assigned to this group are treated with D064, D701, placebo of D012
  Other Names: D064, D701 are consisted of antihypertensive agent.
  Arms: Experimental Group
Drug: D012, placebo of D064, placebo of D701 — Comparator Group Subjects assigned to this group are treated with D012, placebo of D064, placebo of D701
  Other Names: D012 is consisted of antihypertensive agent.
  Arms: Comparator Group

SUMMARY:
Clinical Trial to Evaluate the Efficacy and Safety of D064 and D701 Combination Therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are 19 years old or older.
2. Subjects who have voluntarily decided to participate in this clinical trial and signed ICF.

Exclusion Criteria:

1. Subjects with a history of secondary hypertension or suspected secondary hypertension
2. Subjects who require combination administration of antihypertensive drugs other than clinical trial drugs during the clinical trial participation period
3. Subjects with hypersensitivity or history of clinical trial drugs and similar drugs
4. Subjects who are required to administer a combination of prohibited drugs specified in this plan during the clinical trial participation period
5. Subjects with a history of drug or alcohol abuse or suspected patient within 24 weeks as of the time of screening
6. Subjects who received other clinical trial drugs within 4 weeks of screening visit.
7. Pregnant women, lactating women, or Subjects who do not agree to use appropriate contraception during the clinical trial period and for two weeks after the end of administration of the last clinical trial drug
8. Subjects who are unable to participate in this clinical trial at the discretion of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in MSSBP | 8 weeks after drug administrations
  Compare experimental group with comparator group

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No